CLINICAL TRIAL: NCT06444750
Title: Comparison of the Proteome in ICU Patients in Search for TRALI Biomarkers: A Case-control Study Using Both Retrospective and Prospective Samples
Acronym: CURIE
Status: Not yet recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, A.P.J. Vlaar, Head of department of Intensive Care Medicine, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: CURIE
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Transfusion-Related Acute Lung Injury; ARDS, Human
Keywords: Transfusion-Related Acute Lung Injury; Proteomics; Intensive Care Unit; Critical Ill patients
MeSH Terms: conditions — Transfusion-Related Acute Lung Injury; Respiratory Distress Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- ICU patients who receive a transfusion without lung injury: Purpose: This group is critical for comparing the baseline effects of blood transfusion on the proteome in critically ill patients who do not develop lung injury Following transfusion, providing a control to differentiate between transfusion-related changes in the blood composition and the specific lung injury observed in TRALI. Understanding these changes will help identify biomarkers and mechanisms exclusive to TRALI. Research question: How do transfusion-related proteomic changes manifest in ICU patients who do not develop lung injury after transfusion, and how does this baseline differ from the proteomics of TRALI patients?
  Interventions: Other: Blood sample collection
- ICU patients who receive a transfusion and have indirect ARDS: Purpose: By excluding patients with ARDS due to a pulmonary cause, this group isolates systemic, non-pulmonary factors that trigger lung injury from local pulmonary responses.
  Comparing this with TRALI helps us pinpoint unique biomarkers and understand the role of plasma proteins and various cellular-pathways dealing with systemic inflammation with concomitant lung injury. Research question: What distinct proteomic profiles and cellular pathways in non-pulmonary ARDS are observed in comparison with TRALI?
  Interventions: Other: Blood sample collection
- ICU patients who receive a transfusion and have infectious pneumonia: Purpose: Since both TRALI and pneumonia involve lung injury, understanding the differences in these responses will provide insight into the mechanisms responsible for lung inflammation in TRALI, distinguishing it from the lung inflammation caused by local pulmonary infection.
  Research question: Can we differentiate between the immune and proteomic responses in localized infectious lung injury and transfusion-induced TRALI, exposing how the immune system reacts to an infection versus a transfusion event?
  Interventions: Other: Blood sample collection
- ICU patients without transfusion and with indirect ARDS: Purpose: This group allows us to characterize the proteomic and immunological responses of ARDS independent of transfusion events. This comparison with TRALI aids in the identification of changes solely due to transfusion-induced acute lung injury. Research question: What are the unique blood signatures in indirect ARDS patients when transfusion factors are removed from the equation?
  Interventions: Other: Blood sample collection
- Patients without transfusion and with infectious pneumonia: Purpose: Including this group clarifies the distinction between changes driven by infection and those unique to transfusion. By subtracting the effects of infectious responses, we can confirm that biomarkers are related specifically to TRALI. ABR 86798 CURIE study Version 5,April, 2025 16 of 35 Research question: How do the inflammatory cell and protein responses to localized lung infections compare to those induced by TRALI, ensuring biomarkers identified are specific to transfusion-related injury?
  Interventions: Other: Blood sample collection
- Healthy volunteers: Purpose: The inclusion of healthy volunteers in this study is crucial. They provide a baseline of normal physiological and immunological steady-state composition of the blood, allowing us to identify biomarkers specific to TRALI and the other patient subgroups by accounting for baseline variability. This group serves as a valuable control for confounding factors such as critical illness (for which ICU admission), or pre-existing lung injury or concomitant systemic inflammation including the lung (ARDS), which might otherwise obscure the identification of TRALI-specific changes. This enhances data analysis and provides clarity in distinguishing potentially unique pathophysiologic mechanisms in TRALI.
  Research question:
  What baseline levels of protein, immune, and cellular profiles in healthy individuals differ from those in ICU patients undergoing transfusion, particular in terms of neutrophil activity, Treg function, and overall inflammation
  Interventions: Other: Blood sample collection

INTERVENTIONS:
Other: Blood sample collection — Blood samples of 30 mL will be collected at admission. For the groups that receive a blood transfusion an extra 30 mL blood sample will be collected.
  Other Names: Blood draw

SUMMARY:
Transfusion-related acute lung injury (TRALI) is a severe complication of blood transfusions. After a transfusion, TRALI develops in 0.08-15% of cases depending on the characteristics of the studied population. Due to preventive measures the incidence has decreased. However, the incidence of TRALI is 50-100 times higher in critically ill patients compared to the general hospital population. Since the absolute incidence of respiratory transfusion complications is low and TRALI is under-diagnosed and - reported, to this date is has not been possible to elucidate the exact pathophysiology of TRALI. Consequently, no biomarkers are yet known to detect TRALI. This study aims to identify TRALI biomarkers, gain insight in cellular pathways underlying TRALI development and the role of neutrophils and regulatory T cells, which could enhance transfusion safety.

DETAILED DESCRIPTION:
Objective of the study:

* To identify biomarkers specific for TRALI, thus aiding in future diagnostics of TRALI.
* To investigate the proteome in TRALI patients and thus gain knowledge on TRALI pathophysiology. This knowledge can be used to investigate preventive measures and therapy for TRALI.
* To investigate the role of neutrophils and regulatory T cells in TRALI, which are thought to be essential dysregulated in the in TRALI pathogenesis.

Study design:

Case-control study using retrospective and prospective samples. Samples available from known TRALI patients stored at Sanquin Blood Bank will be compared to samples from intensive care patients with acute respiratory distress syndrome (ARDS), pneumonia, or without lung injury and to samples of healthy volunteers. The treating physician will screen ICU patients for eligibility for one of our groups and asks for permission to be approached by a researcher for informed consent. After obtaining informed consent, patients will be allocated to a group depending on whether they need a transfusion. After admission and informed consent extra blood samples (30ml) will be drawn from patients within 24 hours of arrival.

For Group 1 (patients who receive a transfusion but do not have lung injury), Group 2 (patients who receive a transfusion and have indirect ARDS), and Group 3 (patients who receive a transfusion with pneumonia (local lung injury)) a second tube blood sample (30ml) will be drawn 12 hours after the first transfusion. We will collect two samples (max 60 mL) for this group to analyze the effect of transfusion on the proteome. Together with the clinical data we will search for TRALI biomarkers.

Study population:

Adult intensive care patient who are admitted with:

Pneumonia (without ARDS), indirect ARDS or no pulmonary injury with and wihtout receiving a blood transfusion.

Healthy volunteers obtained through the Sanquin donor system. The TRALI samples that are obtained through hemovigilance at Sanquin (see protocol 4.1).

Primary study parameters/outcome of the study:

The primary endpoint of this study is to identify TRALI-specific biomarkers by comparing plasma proteomic profiles between the following groups: TRALI patients, indirect ARDS patients (with and without transfusion), pneumonia patients (with and without transfusion), and healthy volunteers. To isolate the impact of transfusion on the proteome and differentiate it from TRALI-specific changes, we will also analyze proteomic profiles before and after transfusion in relevant groups. This approach aims to increase the specificity and sensitivity of identified protein biomarkers for accurate TRALI diagnosis and facilitate the development of novel diagnostic assays.

Secundary study parameters/outcome of the study (if applicable):

The secundary outcomes of this study are:

1. Characterizing the TRALI Proteome: we will perform in-depth characterization of the proteome in TRALI patients to gain a comprehensive understanding of the molecular mechanisms underlying TRALI pathophysiology. This analysis aims to uncover potential therapeutic targets and pathways involved in TRALI development.
2. Investigating Neutrophil and Treg responses: we will investigate the phenotype, activation status, and functional responses of neutrophils and Tregs in TRALI patients compared to relevant control groups. This detailed analysis will shed light on the roles of neutrophils and Tregs in TRALI pathogenesis.

ELIGIBILITY:
Inclusion criteria

Patients on the ICU:

1. Without lung injury who received a red blood cell (RBC) or platelet transfusion (PLT).
2. With indirect ARDS with and without a blood transfusion (RBC or PLT);
3. With pneumonia, with and without a blood transfusion (RBC or PLT).

Exclusion criteria

1. "Objection to registration of data for scientific use" as noted in the patient file.
2. Patients in whom it is impossible to obtain blood samples.
3. Patients with massive hemorrhage.
4. Patients with ARDS due to multiple transfusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Samples from twenty TRALI patients are already available at Sanquin Blood Bank. These samples have been collected within 24 hours after TRALI onset. The only clinical data available for these samples is sex and age. This is our study group. As control we will include ICU patients in University Medical Center (UMC):
  * Patients without lung injury receiving a blood transfusion;
  * Patients with indirect ARDS receiving a blood transfusion;
  * Patients with pneumonia receiving a blood transfusion;
  * Patients with indirect ARDS, who do not receive a blood transfusion;
  * Patients with pneumonia who do not receive a blood transfusion;
  * Healthy volunteers recruited through Sanquin's donor system
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Biomarkers for TRALI | From admission to the end of data collection (30 days)
  The primary endpoint of this study is to identify TRALI-specific biomarkers by comparing plasma proteomic profiles between the following groups: TRALI patients, indirect ARDS patients (with and without transfusion), pneumonia patients (with and without transfusion), and healthy volunteers. To isolate the impact of transfusion on the proteome and differentiate it from TRALI-specific changes, we will also analyze proteomic profiles before and after transfusion in relevant groups. This approach aims to increase the specificity and sensitivity of identified protein biomarkers for accurate TRALI diagnosis and facilitate the development of novel diagnostic assays

SECONDARY OUTCOMES:
Characterizing the TRALI proteome | From admission to the end of data collection (30 days)
  We will perform in-depth characterization of the proteome in TRALI patients to gain a comprehensive understanding of the molecular mechanisms underlying TRALI pathophysiology. This analysis aims to uncover potential therapeutic targets and pathways involved in TRALI development.
Investigating Neutrophil and Treg responses | From admission to the end of data collection (30 days)
  We will investigate the phenotype, activation status, and functional responses of neutrophils and Tregs in TRALI patients compared to relevant control groups. This detailed analysis will shed light on the roles of neutrophils and Tregs in TRALI pathogenesis.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Vlaar, Professor, Principal Investigator — Amsterdam UMC